CLINICAL TRIAL: NCT03364114
Title: Interscope Endorotor® Mucosal Resection System With Continued Ablative Therapy In Subjects With Refractory Dysplastic Barrett's Esophagus
Brief Title: Endorotor Resection In Refractory Barrett's Dysplasia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Interscope, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0010
Record Dates: First submitted 2017-11-29; First posted 2017-12-06 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Barrett's Esophagus With Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EndoRotor Resection (Experimental): For the purpose of this study the EndoRotor System is investigationally indicated for use during endoscopic procedures to resect and remove refractory Barrett's esophagus tissue in conjunction with a submucosal saline injection mix using adrenaline and dye. Subjects randomized to the EndoRotor arm will be treated up to 3 times through the 9 month follow-up period to remove gross visible Barrett's.
  Interventions: Device: EndoRotor Mucosal Resection System
- Continued Ablation (Control) (Active Comparator): The investigator shall exercise standard of care for subjects undergoing continued ablative therapies (RFA and/or Cryotherapy). These will constitute the control devices. The investigator will choose the system in this arm. Operation of each system will be done according to the manufacturer's IFU. Subjects randomized to the control arm may be treated up to 3 time through the 9 month follow-up period to remove gross visible Barrett's.
  Interventions: Device: Continued Ablation

INTERVENTIONS:
Device: EndoRotor Mucosal Resection System — The EndoRotor® Endoscopic Mucosal Resection System is an automated mechanical endoscopic mucosal resection system for use in the gastrointestinal tract for benign neoplastic or pre-malignant tissue removal by interventional gastroenterologists and GI surgeons. The EndoRotor® System performs both tissue dissection and resection with a single device through an endoscope's instrument biopsy channel.
  Arms: EndoRotor Resection
Device: Continued Ablation — Continued ablation control shall include either cryotherapy or continued radial frequency ablation.
  Arms: Continued Ablation (Control)

SUMMARY:
The aim of the clinical trial is to evaluate the EndoRotor®'s ability to completely remove areas of Barrett's esophagus considered refractory after 3 failed ablation treatments (Radiofrequency Ablation (RFA) and/or Cryotherapy) or in patients with at least 1 failed ablative procedure (RFA and/or Cryotherapy) and are intolerant to the procedure due to pain, where intolerant is defined as post-dysphagia or odynophagia persisting for 24 hours or greater or requiring narcotic analgesia for a duration of more than 24 hours.

DETAILED DESCRIPTION:
Prospective, multi-center, randomized controlled trial, pivotal, investigational device exemption (IDE) to compare the safety and performance of the EndoRotor® Mucosal Resection System with continued ablative therapy in subjects with refractory Barrett's Esophagus.

The EndoRotor® Endoscopic Mucosal Resection System is an automated mechanical endoscopic mucosal resection system for use in the gastrointestinal tract for benign neoplastic or pre-malignant tissue removal by interventional gastroenterologists and GI surgeons. The EndoRotor® System performs both tissue dissection and resection with a single device through an endoscope's instrument biopsy channel.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are greater than 30 and less than 90 years of age; inclusive of males and females.
2. Subjects with confirmed Barrett's esophagus with dysplasia (low-grade or high-grade) and meeting at least one of the following criteria:

   1. Failed 3 ablative procedures (RFA and/or Cryotherapy).
   2. Failed at least 1 ablative procedure (RFA and/or Cryotherapy) and are intolerant to the procedure due to pain, where intolerant is defined as post-procedure dysphagia or odynophagia persisting for 24 hours or greater or requiring narcotic analgesia for a duration of more than 24 hours.
3. Residual Barrett's length is ≥1 cm and ≤6 cm.
4. No confirmed evidence of esophageal adenocarcinoma (EAC) at the time of therapy.
5. Subject capable of giving informed consent.
6. Subject has a reasonable expectation for prolonged survival (greater than 2 years).
7. Subject can tolerate repeated endoscopic procedures.
8. Absence of strictures refractory to dilation that preclude the passage of the endoscope
9. Patients who were on acid suppression therapy (i.e. PPIs) during the course of failed primary ablative therapy, and who can continue acid suppression therapy for the entire time they are on the clinical study.
10. Subjects with the ability to understand the requirements of the study, who have provided written informed consent, and who are willing and able to return for the required follow-up assessments through 12 months, as indicated.

Exclusion Criteria:

1. Subject unable to give informed consent.
2. Subject is unwilling to return for repeated endoscopies.
3. Confirmed endoscopic and or histologic evidence of EAC at time of therapy.
4. Residual Barrett's longer than 6 cm.
5. Subjects with nodular Barrett's esophagus.
6. Subjects who are on anticoagulant therapy that cannot be discontinued for 5 days before and after the procedure.
7. Subjects with known coagulopathy defined as abnormal prothrombin or partial thromboplastin time.
8. History of esophageal varices
9. LA Grade B, C, or D esophagitis.
10. Esophageal stricture refractory to dilation preventing passage of endoscope or catheter.
11. Any previous esophageal surgery, except fundoplication without complications.
12. Medically uncorrectable hypotension or hypertension.
13. Any condition that in the opinion of the investigator would create an unsafe clinical situation that would not allow the patient to safely undergo an endoscopic procedure (lack of medical clearance).
14. Pregnant or lactating women or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator, and/or are not willing to use reliable contraception for the duration of study participation.
15. Subject has known severe psychiatric disorder, substance abuse, or other reason for being unable to follow trial follow-up instructions.
16. Patient has a known significant concomitant illness with a life expectancy of less than 2 years.
17. Subject is known to be currently enrolled in another investigational trial that could interfere with the endpoint analyses of this trial.

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete removal of refractory Barrett's esophagus | 12 months
  The primary effectiveness endpoint for this study is the complete removal of refractory Barrett's esophagus in no more than three treatments as assessed by a biopsy negative for Barrett's esophagus at the 12 month follow-up visit.
Rate of device- and procedure-related serious adverse events (SAEs) | 12 months
  The primary safety endpoint for this study is the rate of device- and procedure-related serious adverse events (SAEs) for bleeding, perforation, and stricture in the EndoRotor arm will be no greater than that of the continued ablative therapy arm.

SECONDARY OUTCOMES:
Activated Fibroblasts | 12 months
  Percent reduction of activated fibroblasts in the area with Barrett's esophagus that was resected using EndoRotor at initial treatment session through the 12 month follow-up visit as per the histological findings of keyhole technique biopsies. - this point is only assessed in the first 5 EndoRotor subjects
Percent Reduction of Barrett's Esophagus | 12 months
  Percent reduction of Barrett's esophagus that was resected or ablated during the initial treatment session through the 12 month follow-up visit as calculated using the Prague classification measurements of estimated circumference and maximal length.
Post Procedure Pain | 9 months
  Assessment of subject post procedure pain as compared to the control arm by means of a visual analogue pain scale.
  The visual analogue pain scale used for this study allows a patient to record their pain using a scoring system from 0 to 10. Zero representing no pain, 5 representing moderate pain, and 10 representing the worst possible pain. Lower scores represent a better score.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wang, MD, Principal Investigator — The Mayo Clinic
Locations (5):
- United States (2):
  - The Mayo Clinic, Rochester, Minnesota
  - University of Rochester Medical Center, Rochester, New York
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (2):
  - NHS University College Hospital, London
  - Nottingham University Hospitals NHS Trust and University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03364114/Prot_SAP_000.pdf